CLINICAL TRIAL: NCT06980051
Title: The Impact of Virtual Windows on Teachers in Windowless Classrooms
Brief Title: Virtual Windows in a Windowless Classroom
Status: Not yet recruiting | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Jamie Zeitzer, Professor, Stanford University
Other Study IDs: IRB-80880
Record Dates: First submitted 2025-05-09; First posted 2025-05-20 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Mood
Keywords: light; mood

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Teachers: Teachers at The Inspired Community Project in the Bronx NY
  Interventions: Behavioral: Virtual window

INTERVENTIONS:
Behavioral: Virtual window — The virtual window, which displays 24h time-linked outdoor scene on a high-definition video monitor, will be on during working hours for three days each week.

SUMMARY:
The investigators are testing whether the use of virtual windows in a windowless classroom environment improves mood among teachers.

DETAILED DESCRIPTION:
Teachers at The Inspired Community Project in the Bronx NY will be exposed to the virtual windows three days per week and the windows will be turned off two days per week. This will last for up to three months. Mood will be tracked.

ELIGIBILITY:
Inclusion Criteria:

* Teacher at The Inspired Community Project, Bronx NY

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Teachers at The Inspired Community Project, Bronx NY
Sampling Method: Non-Probability Sample
Enrollment: 14 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-01-15 (Estimated)

PRIMARY OUTCOMES:
Mood | From enrollment until the end of three months
  Daily Short Messaging Service (SMS)-based assessment of mood

IPD SHARING:
Plan to Share IPD: Yes
De-identified mood data and the associated data concerning whether the virtual window was active will be placed in a public data repository.
Time Frame: The data will be made available by January 5, 2026. There is no end date.
Access Criteria: There is no restriction on access.
URL: https://datadryad.org/